CLINICAL TRIAL: NCT05697289
Title: Satisfaction of HIV-infected Patients Treated With Cabotegravir-rilpivirine Injectable Dual Therapy
Acronym: CABORI
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP221099
Record Dates: First submitted 2022-12-07; First posted 2023-01-25 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2022-01

CONDITIONS: HIV Infections
Keywords: hiv; Cabotegravir-rilpivirine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: satisfaction survey — Non-comparative longitudinal observational study over 12 months conducted during usual follow-up of patients living with HIV-1 and having changed treatment for an injectable dual therapy with prolonged release cabotegravir-rilpivirine. Decision to change treatment and follow-up of patients are part of routine care. Study is proposed after the doctor has taken the decision to modify treatment, the patient has accepted and injectable dual therapy is prescribed. It is based on self-questionnaires to collect patient perceptions (Patient-Reported Outcomes) and clinical and biological data collected routinely at inclusion and during follow-up visits.

SUMMARY:
Question arises as to whether this new treatment "Cabotegravir-rilpivirineactually" improves patient satisfaction and whether it is well suited to everyone, especially those with a history of irregular follow-up. Also, inconvenience of two intramuscular injections every two months and constraint of care organization could represent a barrier to treatment for some patients.

DETAILED DESCRIPTION:
Cabotegravir-rilpivirine prolonged-release injectable dual therapy antiretroviral treatment recently obtained marketing authorization in France to treat human immunodeficiency virus (HIV) infection. It would meet the demand of patients for less frequent treatment to overcome constraints associated with daily drug intake such as stigma due to HIV, weight of daily pill recalling disease or difficulties in compliance. This authorization follows the results of FLAIR and ATLAS phase III clinical trials, which showed non-inferiority of monthly injectable treatment in terms of virological control compared to conventional oral triple therapy. 1-4 ATLAS-trial 2M showed non-inferiority of injectable treatment every two months compared to every month.5 Main risk factors for virological failure highlighted were a low residual plasma concentration of rilpivirine, viral subtype A1/A6, existence of archived resistance mutations to rilpivirine and obesity (BMI > 30 kg/ m²).6 Discontinuation rate of injectable treatment at one year was 9% in FLAIR trial and 8% in ATLAS versus 8% and 6% respectively for control group under oral treatment. Most treatment discontinuations were due to adverse effects.

Most commonly reported adverse reactions were injection site reactions (up to 84%), headache (up to 12%) and fever (10%). In these studies, patient satisfaction was assessed through multiple scales or questionnaires. Results of these evaluations did not make it possible to conclude on the impact of injectable treatment on patients quality of life.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected patient
* Patient over 18 years of age
* Patient for whom dual injectable sustained-release cabotegravir-rilpivirine therapy is implemented according to the decision of the referring physician in the context of care.
* Patient who understands, reads and writes French well

Exclusion Criteria:

* Patient opposing to participate in the study.
* Patient subject to legal protection measures (guardianship, curatorship or safeguard of justice)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients living with HIV-1 and having changed treatment for an injectable dual therapy with prolonged release cabotegravir-rilpivirine.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
treatment satisfaction in people living with HIV | 12 months
  Change in human immunodeficiency virus Treatment Satisfaction Questionnaire (HIVTSQ12) status version score between conventional oral tri-therapy and after one year of intramuscular injectable bi-therapy.

SECONDARY OUTCOMES:
Proportion of patients who stopped treatment, median duration of treatment and reason for stopping. | 12 months
  duration of treatment and reason for discontinuation.
Satisfaction : Change in human immunodeficiency virus Treatment Satisfaction Questionnaire (HIVTSQ12) status score between conventional oral triple therapy D0 and after 6 months of intramuscular dual therapy M6, | 12 months
  adherence to treatment and compliance with the injection schedule
Compliance: number of patients who received an injection more than 7 days after the scheduled date | 12 months
  patients perceptions of cabotegravir-rilpivirine injectable dual therapy.
CD4 cells count | 12 months
  Immuno-virological control: CD4 count